CLINICAL TRIAL: NCT00384007
Title: A Randomized Trial Comparing SpineJet® Hydrodiscectomy to Open Lumbar Microdiscectomy for Treatment of Lumbar Radiculopathy Due to Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pinnacle Pain Medicine (Industry)
Collaborators: HydroCision, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-SJ-1001
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Disc Herniation With Radiculopathy
Keywords: back pain; herniated disc; leg pain; pinched nerves; sciatica; radiculopathy
MeSH Terms: conditions — Back Pain; Intervertebral Disc Displacement; Sciatica; Radiculopathy

INTERVENTIONS:
Procedure: Hydrodiscectomy with Spinejet

SUMMARY:
The purpose of this study is to compare a standard surgical procedure, open surgical microdiscectomy, used primarily to relieve leg pain and repair disc herniation to a newer surgical procedure, hydrodiscectomy with Spinejet®. The study will examine how well each procedure reduces subject pain and disability over a one-year period. Magnetic resonance imaging (MRI-use of a magnetic field to produce an image) of the lower spinal column taken before and after surgery will also be looked at to determine what physical changes have taken place over the course of a year. Subjects enrolled in this study will also be asked to keep track of their medical expenses related to treating their back pain to see if the surgeries being compared reduce out of pocket expenses.

DETAILED DESCRIPTION:
This is a randomized multi-clinic study supported by HydroCision, Inc. to compare open lumbar microdiscectomy to percutaneous lumbar discectomy with Spinejet® for patients with contained or small extruded disc herniation with nerve root contact and concordant radiculopathy. Initially this pilot study will enroll 20 patients over 6 months after which statistical analysis will be performed to evaluate the merit of continuing the study. Patients will be randomized in a 1:1 ratio. If a study participant has been randomized to receive open lumbar microdiscectomy a referral to a neurosurgeon will be made for the patient. All patients participating in study must be screened, meet all study inclusion/exclusion criteria and sign informed consent and HIPAA forms prior to any research participation. Once randomization to receive either hydrodiscectomy with Spinejet® or open lumbar microdiscectomy has occurred study participants will be evaluated within two weeks of scheduled procedure. If a patient randomized to either group refuses the proposed treatment plan, they will be removed as a study participant. At the pre-op visit patient demographics, history, healthcare coverage, duration of symptoms, concomitant medications, level of HNP, MRI, Visual Analog Scale (VAS), Beck's Inventory Depression (BID) scale and the Oswestry Disability Index (ODI) score as well as Lumbar Spine Outcomes questionnaire (LSOQ) will be collected. At the time of surgery all patients will have discography at the surgical level with 2cc Isovue contrast injected at 0.04cc/sec. Evidence of epidural extravasation would exclude a patient from further study participation. At the completion of the procedure device run time and length of procedure will be recorded. Post-operative patients will return to clinic for 5 follow-up visits, being evaluated at 1 week, 1 month, 3 month, 6 month and 12 month intervals. Blinded observers will record sensory deficits to touch, pain, temperature, motor strength of major muscle groups, patient reflexes(0-4 scale),SLR (degrees in prone position) analgesics dose and frequency. Patients will also complete VAS, BID, LSOQ, and ODI score calculated at each follow-up visit. MRIs will be performed at 1month follow-up visit for patients having hydrodiscectomy with all study participants having an MRI at the 12 month visit. MRIs will be read by a radiologist blinded to study procedure to determine type, size of protrusion and nerve root contact. Patients will be asked about any adverse events, changes in medications, or any health concerns at each follow-visit. Over the course of the study patients will also be asked to keep a study-specific log of expenses incurred due to back pain. Physicians and patients participating in the study will each be paid $50.00 per study visit for a maximum of $300.00. Imaging studies and hydrodiscectomy procedures will be provided to the patient at no charge other than copay/deductibles if paid by a third party payer.

ELIGIBILITY:
Inclusion Criteria:

* Patient ages 18-75, both sexes
* Posterolateral single lumbar contained disc herniation, any level, up to 1/3 of spinal canal sagittal diameter, concordant radicular pain +/- back pain, and MRI confirmed nerve root contact/compression
* Failed trial of at least one NSAID within 6 months
* Failed at least 2 weeks physical therapy within 6 months
* Failed at least 2 epidural steroid injection (ESIs), no less than 2 weeks apart within 6 months
* Initial or recurrent episode of radiculitis
* Willingness to sign IRB-approved consent

Exclusion Criteria:

* Strength < 4/5 in major muscle group of ipsilateral lower extremity
* Large extruded or sequestered HNP
* Greater than mild central canal, lateral recess, or neuroforamenal stenosis
* Previous surgery at affected level
* Other level lumbar HNP on affected side
* Significant (>50%) loss of disc height compared to the adjacent higher level
* Local infection at needle insertion site
* Epidural extravasation on discography
* Pregnancy
* ASA status IV/V
* Diseases transmitted by blood
* Any illness, condition, or medication that would make a patient unsuitable for a surgical procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Pain reduction

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Wasserman, M.D., Principal Investigator — Pinnacle Pain Medicine
Locations (1):
- Pinnacle Anesthesia Consultants, P.A. d.b.a. Pinnacle Pain Medicine, Dallas, Texas, United States